CLINICAL TRIAL: NCT02291874
Title: Postmarketing Clinical Study of Ipragliflozin - Long-term Study in Combination With GLP-1 Receptor Agonists in Patients With Type 2 Diabetes Mellitus
Brief Title: Post-Marketing Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of Ipragliflozin in Combination With GLP-1 Receptor Agonists in Japanese Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1941-CL-0132
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Ipragliflozin; GLP-1 receptor agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipragliflozin group (Experimental): Ipragliflozin treatment
  Interventions: Drug: Ipragliflozin

INTERVENTIONS:
Drug: Ipragliflozin — oral
  Other Names: Suglat tablet; ASP1941

SUMMARY:
Purpose of this study is to evaluate the Long-term Safety, Tolerability, and Efficacy of Ipragliflozin in Combination with GLP-1 Receptor Agonists in Japanese Patients with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control with GLP-1 Receptor Agonists.

DETAILED DESCRIPTION:
This is a multicenter, open-label study in patients with T2DM who have inadequate glycemic control with GLP-1 receptor agonists for at least 6 weeks prior to Visit 1 (Week -6).

Patients on monotherapy with Victoza® or on combination therapy with GLP-1 receptor agonists and sulfonylurea (SU) are eligible. Patients on combination therapy with GLP-1 receptor agonists and non-SU hypoglycemic agents can also be included; however, these patients must undergo washout of the non-SU hypoglycemic agents administered with GLP-1 receptor agonists.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a diagnosis of T2DM that was determined at least 12 weeks (84 days) before providing informed consent.
* The subject has been receiving the same GLP-1 receptor agonist at a fixed dose and mode of administration for at least 6 weeks (42 days) prior to Visit 1.
* If on therapy with a concomitant SU, the subject has been receiving the same SU at a fixed dose and mode of administration for at least 6 weeks (42 days) prior to Visit 1.
* The subject has HbA1c levels of ≥7.5% but ≤10.5% at Visit 2, and the difference in HbA1c levels between Visit 1 and Visit 2 is within ±1.0%.
* The subject has a BMI of ≥20.0 kg/m2 but ≤45.0 kg/m2 at Visit 2.
* If on therapy with a concomitant SU, the subject has fasting plasma glucose levels of ≥126 mg/dL at Visit 2.

Exclusion Criteria:

* The subject has T1DM.
* The subject has symptoms of dysuria, anuria, oliguria, or urinary retention.
* The subject has proliferative retinopathy.
* The subject has a history of clinically significant renal diseases such as renovascular occlusive disease, nephrectomy, or renal transplant.
* The subject has a history of pancreatitis.
* The subject has a history of recurrent urinary tract infections (≥3 episodes within 24 weeks before providing informed consent).
* The subject has a symptomatic urinary tract infection or symptomatic genital infection.
* The subject has a chronic disease that requires the continuous use of adrenocortical steroids and immunosuppressants (oral, injectable, or inhalational medications).
* The subject has a history of cerebral vascular attack, unstable angina, myocardial infarction, vascular intervention, or serious heart disease (NYHA Class III-IV) within 1 year (52 weeks) prior to Visit 1, or the subject has heart disease or cerebral vascular disease that, as per the judgment of the investigator or sub-investigator, may interfere with the treatment with ipragliflozin or safety evaluation of this study.
* The subject has an unstable psychiatric disorder.
* The subject is a female who is currently pregnant or lactating or could be pregnant.
* The subject is unable or unwilling to practice an appropriate contraception method during the study.
* The subject has severe infection, perioperative or serious trauma.
* The subject has drug addiction or abuses alcohol.
* The subject has a history of malignant tumors (except when he/she has been free from treatment for at least 5 years before providing informed consent and is not considered to have any recurrence).
* The subject has a history of allergy to ipragliflozin or similar drugs that have an SGLT2 inhibitory action.
* The subject has participated in a clinical study of an investigational product or medical device or post-marketing study within 12 weeks (84 days) before providing informed consent or is currently participating in any of these studies.
* The subject is unable or unwilling, or does not agree, to comply with the study requirements, including the hospital visits, dose instructions, and the subject's responsibilities.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Fasting plasma glucose | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week

SECONDARY OUTCOMES:
Fasting serum insulin | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Serum glucagon | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Serum glycoalbumin | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Serum leptin | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Serum adiponectin | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Body weight | 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Waist circumference | at 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52-week
Self-measured blood glucose | at 0, 20, 52-week
  Subjects measure blood glucose 7 times a day on any 3 days in a week before each scheduled visit and record the results in the patient diary
Adverse events (AEs), vital signs, and laboratory tests | All treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Ishihara H, Yamaguchi S, Nakao I, Sakatani T. Ipragliflozin Add-on Therapy to a GLP-1 Receptor Agonist in Japanese Patients with Type 2 Diabetes (AGATE): A 52-Week Open-Label Study. Diabetes Ther. 2018 Aug;9(4):1549-1567. doi: 10.1007/s13300-018-0455-8. Epub 2018 Jun 20. PMID 29926400
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=220